CLINICAL TRIAL: NCT06978491
Title: Evaluation of the Effect of Postoperative Analgesia Techniques on Obstetric Recovery Quality With ObsQoR-10
Brief Title: Evaluation of the Effect of Postoperative Analgesia Techniques With ObsQoR-10
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Meryem Onay, Associate professor, Anesthesiologist, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESOGU 6
Record Dates: First submitted 2025-05-11; First posted 2025-05-18 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-04

CONDITIONS: Pain, Postoperative; Postoperative Complications
Keywords: cesarean section; postoperative analgesia; Quality of recovery
MeSH Terms: conditions — Pain, Postoperative; Postoperative Complications | interventions — Sensitivity Training Groups

STUDY DESIGN:
Intervention Model Description: Group C: spinal anesthesia.
  Group T: spinal anesthesia and at the end of the surgery, 0.25% bupivacaine and 20 ml of local anesthetic will be applied bilaterally between the transversus abdominis and internal oblique muscle.
  Group W (wound infiltration) : spinal anesthesia and at the end of the surgery, 0.25% bupivacaine and 20 ml of local anesthetic will be applied to the wound site.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group C (Control) (Active Comparator): spinal anesthesia.
  Interventions: Other: Group C
- Group T (Transversus Abdominis Plane Block) (Active Comparator): The operation will be performed under spinal anesthesia and at the end of the operation, 20 ml of 0.25% bupivacaine will be applied bilaterally between the transverse abdominis muscle and the internal oblique muscle.
  Interventions: Other: Group T
- Group W (Wound Infıltration) (Active Comparator): The operation will be performed under spinal anesthesia and at the end of the operation, 20 ml of 0.25% bupivacaine will be applied wound infiltration
  Interventions: Other: Group W

INTERVENTIONS:
Other: Group C — Spinal anesthesia.
  Other Names: Control
  Arms: Group C (Control)
Other: Group T — spinal anesthesia and at the end of the surgery, 20 ml 0.25% bupivacaine will be applied bilaterally between the transversus abdominis and internal oblique muscle.
  Other Names: Transversus Abdominis Plane Block
  Arms: Group T (Transversus Abdominis Plane Block)
Other: Group W — spinal anesthesia and at the end of the surgery, 20 ml 0.25% bupivacaine will be applied to the wound site.
  Other Names: Wound Infıltration
  Arms: Group W (Wound Infıltration)

SUMMARY:
The primary objective of this study is to evaluate the effects of postoperative analgesia techniques-transversus abdominis plane (TAP) block and wound infiltration-on recovery in patients undergoing elective cesarean section, using the Obstetric Quality of Recovery-10 (ObsQoR-10) questionnaire. The secondary objective is to assess pain scores, analgesic consumption, and adverse effects such as nausea, vomiting, and pruritus within the first 24 hours postoperatively.

DETAILED DESCRIPTION:
The patients will be divided into 3 groups as Group T (transversus abdominis plane block), Group W (wound infiltration) and Group K (control). All of them will be given spinal anesthesia in sitting position.Group C will receive spinal anesthesia. In Group T (Transversus abdominis plane block) cases, in addition to spinal anesthesia at the end of the surgery, 20 ml of 0.25% bupivacaine will be applied bilaterally between the transversus abdominis muscle and the internal oblique muscle. Group WI (wound infiltration) will be administered 20 ml 0.25% bupivacaine to the wound area in addition to spinal anesthesia at the end of the surgery.Numerical pain scores (NRS Resting and Movement), heart rate, mean arterial pressure, peripheral oxygen saturation, analgesic consumption, nausea and vomiting score, pruritus, Ramsey sedation scale and other postoperative complications will be recorded at the 2nd hour, 6th hour, 12th hour and 24th hour postoperatively .Obstetric Quality of Recovery -ObsQoR-10 questionnaire will be applied to the patients at the end of 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Term obstetric patients aged 18-50 years who underwent elective cesarean section under spinal anesthesia and applied regional anesthesia techniques such as TAP and wound infiltration.

Exclusion Criteria:

* Refuse to participate in the study
* Patients who have undergone general anesthesia
* Patients requiring emergency cesarean section.
* Mental status disorders
* Known bleeding and/or coagulation disorders
* Infection at injection site

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 75 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-05 (Estimated)

PRIMARY OUTCOMES:
Obstetric Quality of Recovery-10 | At postoperative 24th hours
  The ObsQoR-10 questionnaire consists of 10 questions that assess the patient-reported quality of recovery in obstetric patients' postoperative period using an 11-point scale (0 = strongly negative; 10 = strongly positive) that points to a minimum score of 0 (worst possible recovery) and a maximum score of 100 (best possible recovery).

SECONDARY OUTCOMES:
Postoperative pain score, analgesic consumption | At postoperative 24 hours (0, 2, 6,12,24)
  Numeric rating scale pain from 0 (no pain) to 10 (worst pain).

CONTACTS AND LOCATIONS:
Overall Officials: Meryem Onay, Principal Investigator — Eskisehir Osmangazi University Faculty Of Medıcıne
Locations (1):
- Eskisehir Osmangazi Universıty Faculty of Medicine, Eskişehir, Eski̇şehi̇r, Turkey (Türkiye)

REFERENCES:
- [Background] Roofthooft E, Joshi GP, Rawal N, Van de Velde M; PROSPECT Working Group* of the European Society of Regional Anaesthesia and Pain Therapy and supported by the Obstetric Anaesthetists' Association. PROSPECT guideline for elective caesarean section: updated systematic review and procedure-specific postoperative pain management recommendations. Anaesthesia. 2021 May;76(5):665-680. doi: 10.1111/anae.15339. Epub 2020 Dec 28. PMID 33370462
- [Background] Nasir F, Sohail I, Sadiq H, Habib M. Local Wound Infiltration with Ropivacaine for Postoperative Pain Control in Caesarean Section. Cureus. 2019 Sep 5;11(9):e5572. doi: 10.7759/cureus.5572. PMID 31695991
- [Background] Riemma G, Schiattarella A, Cianci S, La Verde M, Morlando M, Sisti G, Esposito I, Della Corte L, Sansone P, De Franciscis P. Transversus abdominis plane block versus wound infiltration for post-cesarean section analgesia: A systematic review and meta-analysis of randomized controlled trials. Int J Gynaecol Obstet. 2021 Jun;153(3):383-392. doi: 10.1002/ijgo.13563. Epub 2021 Feb 11. PMID 33368204
- [Background] Sultan P, Kormendy F, Nishimura S, Carvalho B, Guo N, Papageorgiou C. Comparison of spontaneous versus operative vaginal delivery using Obstetric Quality of Recovery-10 (ObsQoR-10): An observational cohort study. J Clin Anesth. 2020 Aug;63:109781. doi: 10.1016/j.jclinane.2020.109781. Epub 2020 Mar 20. PMID 32203873